CLINICAL TRIAL: NCT06390046
Title: Comparison of Total Intravenous Anesthesia and Inhalational Anesthesia in Opioid-Free Anesthesia for Bariatric Surgery: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, PHD MD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072.6120.135.2023
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-04

CONDITIONS: Analgesics, Opioid; Anesthesia; Adverse Effect

STUDY DESIGN:
Intervention Model Description: The study group will be male and female patients, ASA II or III, over 18 years of age and under 75 years of age. Each patient will undergo abdominal (bariatric) surgery.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA (Active Comparator): total intravenously anesthetized (infusion of Propofol, Ketamine, Lignocaine and Dexmedetomidine)
  Interventions: Drug: TIVA versus Inhalation
- Inhalation agent (Experimental): combined general anesthesia (infusion of Ketamine, Lignocaine and Dexmedetomidine and inhalation of Sevoflurane)
  Interventions: Drug: TIVA versus Inhalation

INTERVENTIONS:
Drug: TIVA versus Inhalation — comparing TIVA with genera anesthesia with inhalation agent

SUMMARY:
Total intravenous general anesthesia and combined general anesthesia are recognized methods used during anesthesia. They allow you to effectively control pain and reduce the number of complications associated with taking large doses of opioid drugs. It should be emphasized that both methods of anesthesia are currently approved for use in routine anesthetic practice, and only the experience, knowledge and preferences of the anesthesiologist determine which technique will be used in a given patient. Both techniques are used in everyday anesthetic practice, but there is no conclusive scientific data confirming the superiority of either method in patients undergoing bariatric surgery, therefore currently only the individual experience, knowledge and preferences of the anesthesiologist determines which technique will be used in a given patient.

DETAILED DESCRIPTION:
Patients undergoing bariatric surgery were randomly divided into two groups: one under complete intravenous anesthesia (infusion of Propofol, Ketamine, Lignocaine and Dexmedetomidine) and the other group under combined general anesthesia (infusion of Ketamine, Lignocaine and Dexmedetomidine and inhalation of Sevoflurane). In the postoperative period, all patients will receive Oxycodone NCA or in the form of oral tablets [naloxone (naloxone hydrochloride) + oxycodone (oxycodone hydrochloride)] and coanalgesics in the form of Paracetamol, Dexac, and Metamizol. Both methods of anesthesia are commonly used and used during bariatric and other surgical procedures. It should be emphasized once again that the above-mentioned all drugs are approved for routine use during anesthesia of patients, including obese patients, and our intervention only involves the use of a specific regimen from among those routinely available. The choice of anesthesia method depends on the anesthesiologist. During the study, we want to randomize patients into two groups: one will be anesthetized using a completely intravenous method, the other will be anesthetized using an inhalation anesthetic. In the postoperative period, patients will have their pain level assessed using the NRS scale 1, 2, 6, 12 and 24 hours after the procedure.

This study aimed to compare TIVA (propofol plus non-opioid adjuncts) with a sevoflurane-based anesthesia protocol, both incorporating OFA principles with lidocaine, ketamine, and dexmedetomidine infusions, in patients undergoing laparoscopic bariatric surgery. We hypothesized that both regimens would provide effective analgesia and recovery, with differences in recovery characteristics and postoperative nausea profiles. Moreover, we intended to evaluate whether a sevoflurane-based approach could match the clinical benefits of TIVA while aligning with current ecological and sustainability priorities in anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years who underwent laparoscopic bariatric surgery

Exclusion Criteria:

Patients with a history of allergic reactions to drugs Patients with a history of drug addiction Patients with chronic pain who require analgesics History of hospitalization for psychiatric disorders Preoperative pulse oximetry (SpO2) < 95 % bradycardia (HR<50bpm), hypotension, atrioventricular block, intraventricular or sinus block Blood clotting disorders Pregnant/lactating women Cognitive impairment Unable to read consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
presence of PONV in postoperative period | 1 day
  The incidence of postoperative nausea and vomiting (PONV) within the first 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative recovery parameters | 1 day
  the measures of return of gastrointestinal function such as volume of oral fluids consumed
Opioid consumption | 1 day
  Postoperative pain levels at 1, 2, 6, 12, and 24 hours were assessed by NRS

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided